CLINICAL TRIAL: NCT04577287
Title: The Effects of Anodal and Cathodal Transcranial Direct Current Stimulation Combined With Conventional Physical Therapy in Patients With Acute Stroke
Brief Title: The Effects of Anodal and Cathodal tDCS Combined With Conventional Physical Therapy in Patients With Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: SI-2842019
Record Dates: First submitted 2020-10-01; First posted 2020-10-06 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cathodal tDCS & PT (Experimental): Cathodal transcranial direct current stimulation (tDCS) will be applied for 20 mins before conventional physical therapy (about 1 hour). Cathode on the on the motor area (M1) of the affected hemisphere, anode on the supraorbital area of the unaffect hemisphere.Current intensity is fixed at 1.5 mA and current will flow continuously. Physical therapist will give an intervention program base on the same basic conventional physical therapy treatment. The scope of intervention is administered to improve motor functions and cerebral hemodynamic .
  Interventions: Device: Transcranial direct current stimulation
- Anodal-tDCS & PT (Experimental): Anodal transcranial direct current stimulation (tDCS) will be applied for 20 mins before conventional physical therapy (about 1 hours). Anode on the motor are (M1) of the affected hemisphere, and cathodal on the supraorbital area of unaffected hemisphere. Current intensity is fixed at 1.5 mA and current will flow continuously. Physical therapist will give an intervention program base on the same basic conventional physical therapy treatment. The scope of intervention is administered to improve motor functions and cerebral hemodynamic .
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Cathodal/Anodal tDCS will be applied in 1.5 mA, 20 mins before conventional physical therapy for 5 days. All experiments will be performed in random order for each subject.

SUMMARY:
The objective of the study is thus to compare the effects 5 consecutive sessions of anodal and cathodal tDCS combined with conventional physical therapy on upper and lower limb motor performance in acute stroke at immediate, and 1-month followup.

DETAILED DESCRIPTION:
Stroke is a major cause of long-term disability in stroke survivors that related with motor impairment. After stroke, the cortical excitability of ipsilesional hemisphere is decreased; in contrast, the cortical excitability of contralesional hemisphere is increased. Conventional physical therapy is beneficial to motor recovery, but early rehabilitation was not always help the patients get full recovery. tDCS is an adjuvant tools which deliver weak direct current through scalp to promote motor recovery in stroke rehabilitation. The anodal-tDCS increases cortical excitability, while the cathodal-tDCS decreases cortical excitability. Previous studies demonstrated that both monocephalic techniques of tDCS can improve motor function in chronic, subacute, and acute phase, but it is still inconclusive that which monocephalic montages had better effect, especially in acute phase. There are several studies supported the benefits of monocephalic tDCS combined with rehabilitation programs on upper and lower limbs motor function in acute stroke. However, there is no evidence that directly compared the effect of monocephalic tDCS in acute stroke patients. The objective of the study is to compare the effects of anodal and cathodal tDCS combined with conventional physical therapy for 5 sessions on motor performance in acute stroke at immediate, and 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke patients who have aged between 18 and 75 years
2. Having a first ever-ischemic stroke that are confirmed by MRI/CT scan
3. Post stroke onset 2-10 days
4. Be able to follow command
5. Be able to walk with or without assistive device (Modified Ranking Scale ≤ 4)
6. Free of any neurological antecedent or unstable condition (such as epilepsy) or cancer.
7. Be able to initiate the upper limb movement

Exclusion Criteria:

1. Recurrent stroke
2. National Institute of Health Stroke Scale ≥ 20 points
3. Presence of intracranial metal implantation, cochlear implant, or cardiac pacemaker
4. Having excessive pain in any joint of the lower limb (numerical pain rating score > 4/10)
5. Having an open wound or wound infraction on scalp
6. Having neglect or psychological diseases (such as schizophrenia, major depression)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 20 minutes
  gold standard and widely used tool to assess sensorimotor in stroke. The item from upper limb and lower limb section will be used. The items are rated on a 3-point ordinal scale as follows: 0 = unable to perform; 1 = partial ability to perform; and 2 = near normal ability to perform.
Wolf Motor Function Test | 5 minutes
  The participants will be asked to perform 2 items that consist of reaching a can and reaching a pen because two tasks is the most common reaching task of hand functions in daily living activities.
Five Times Sit to Stand Test | 5 minutes
  Subjects will sits on the chair and place their back against the chair. Timing will begin at "GO", the subjects will be asked to walk 3m, turn, walk back, and sit down. The stopwatch stops when the patient's buttocks touch the seat.
Time-up and go test | 5 minutes
  The TUG test is a commonly used screening tool to measure basic mobility correlating to dynamic balance. Start from sitting, stand up, walk 3 meters, turn around, walk back 3 meters and sit down. Timed to complete the task represent the body transfer and gait performance
Muscle strength | 10 minutes
  The strength of UE (shoulder flexor, shoulder extensor, elbow extensor, wrist extensor) and LE (hip extensor, hip flexor, knee extensor and ankle dorsiflexor) will be assessed by hand-held dynamometer

SECONDARY OUTCOMES:
Hemodynamic response (VMR%) | 15 minutes
  cerebral blood flow velocity (CBFV), cerebral vasomotor reactivity (VMR) that is the capability of cerebral small vessels to respond to a stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — MU
Locations (1):
- Faculty ofPhysical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No